CLINICAL TRIAL: NCT03697837
Title: Cognitive-Behavioral Therapy for Disruptive Behavior in Children and Adolescents
Brief Title: Digital Parent Training for Disruptive Behaviors in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0102012121-E; 18-004680 (Other Grant/Funding Number: AACAP- Elaine Schlosser Lewis Fund)
Record Dates: First submitted 2018-09-25; First posted 2018-10-05 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Disruptive Behavior; Aggression Childhood; Anger; Non-Compliance, Patient; Irritable Mood
MeSH Terms: conditions — Problem Behavior; Patient Compliance

STUDY DESIGN:
Intervention Model Description: Open feasibility trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parent Management Training (Experimental): Parents will receive a web-based parenting intervention for tantrums and disruptive behavior in young children
  Interventions: Behavioral: Parent Management Training

INTERVENTIONS:
Behavioral: Parent Management Training — The online digital parent training (DPT) program consists of 8 self-guided courses that take approximately 10 minutes to complete and include text and animated parent-child simulations. The courses are designed to closely parallel the content of existing evidence-based parent management training approaches that exist in numerous parenting books.
  Other Names: Digitally-delivered Parent Management Training; PMT

SUMMARY:
This is an open pilot trial of web-based parent training for tantrums and disruptive behavior in children. Parents will be asked to complete a battery of tests to assess their children' behaviors before and after the intervention. Children will undergo a psychiatric evaluation as part of screening. The intervention will be delivered online via an app over a period of 6 weeks. It consists of 8 self-guided courses that take approximately 10 minutes to complete and include text and animated parent-child simulations. Parents will also complete 3 one-hour videoconferencing sessions with a study clinician. During the intervention, parents will be taught various strategies for managing situations that can be anger provoking for their child. This study is conducted to examine whether a digitally-delivered version of parent-management training can be used to reduce behavioral problems including anger outbursts, irritability, aggression and noncompliance.

ELIGIBILITY:
Inclusion Criteria:

* Parents have access to a mobile device and/or computer device
* Parents speak English as native language
* Families agree not to initiate new mental health treatments for the duration of this study.
* Child meets diagnostic criteria for one of the Disruptive Behavior Disorders
* Affective Reactivity Index parent-report score is above 3.6, which is the mean for children with severe irritability
* Lives within driving distance from New Haven, CT

Exclusion Criteria:

* Parents have previously received parent-training by a licensed provider.
* Untreated medical or psychiatric disorder that requires immediate intervention
* Child is non-verbal or minimally verbal

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Feasibility measured by Program completion | Endpoint- Week 6
  Measured by completion of 80% or more of the modules
Feasibility measured by Attendance | Endpoint- Week 6
  Attendance to two of the three videoconferencing sessions
Acceptability measured by Patient Satisfaction Questionnaires | Endpoint- Week 6
  15-item scale measuring satisfaction of participants with clinical intervention

SECONDARY OUTCOMES:
Disruptive Behavior Rating Scale | Baseline (Week 0) and End-point (Week 6)
  16-item rating scale used to assess inattention, hyperactivity-impulsivity, and oppositional defiant behavior among school-aged children. It includes two 8 question subscales, one of which assesses the frequency of these constructs while the other assesses the interference of these constructs in different parts of the child's life. Each item is graded between 0-3 so that each sub-scale has a maximum score of 24 and a minimum score of 0 with a total range of 24. The two subscales are not combined in any way. Higher values are a worse outcome as they either represent a greater frequency or interference (depending on the sub-scale).
MAP-DB- Multidimensional Assessment of Preschool Disruptive Behavior | Baseline (Week 0) and End-point (Week 6)
  A developmentally sensitive questionnaire that includes ~74 items, to assess frequency of temper loss in terms of tantrum features and anger regulation in preschool-aged children. Will perform a preliminary evaluation of intervention effectiveness by assessing change in pre-post scores. Each item is rated on a 6-point likert scale ranging between "never" to "many times each day". The scoring system for this measure is not published, but the authors of this novel tool have agreed to assist in the scoring of this scale.
SNAP-Swanson, Nolan and Pelham Questionnaire (SNAP) | Baseline (Week 0) and Endpoint (Week 6)
  Parent and teacher questionnaires with 18 scored items. Items 1-9 assess inattention in children, while items 11-19 assess hyperactivity in children. Each item ranges between 0-3. Items 10 and 20 are not scored. The higher the score, the worse the outcome as the higher scores reflect greater frequency in the child's inattention or hyperactivity. The two sub-scales are not combined.
CBCL - Child Behavior Checklist | Baseline (Week 0) and Endpoint (Week 6)
  The Child Behavior Checklist is a parent rating of child psychopathology that has factor-analytically derived scales of anxiety, depression, and disruptive behavior. It includes 7 general questions about the child's preferences and activities, and 113 items to assess childhood behavior. We will use it to obtain a more detailed characterization of psychopathology in children.
ARI-Affective Reactivity Index | Screening (Week 0) and Endpoint (Week 6)
  ARI is a 7-item measure of irritability in children and adolescents. Items are rated between 0-2, except for the last item (Number 7) which is not used for scoring. The scale has a minimum score of 0 and a maximum score of 12. An "Affective Reactivity Index Average Score" will be calculated, which is the total score divided by 6. The higher the score, the worse the outcome as this represents greater problems related to irritability. There are no subscales in this measure.

CONTACTS AND LOCATIONS:
Overall Officials: Denis G Sukhodolsky, Ph.D., Principal Investigator — Yale University; Andrea Diaz Stransky, M.D., Principal Investigator — Yale University
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Diaz-Stransky A, Rowley S, Zecher E, Grodberg D, Sukhodolsky DG. Tantrum Tool: Development and Open Pilot Study of Online Parent Training for Irritability and Disruptive Behavior. J Child Adolesc Psychopharmacol. 2020 Nov;30(9):558-566. doi: 10.1089/cap.2020.0089. Epub 2020 Oct 9. PMID 33035067
- See also: Web-based platform for digitally delivered intervention — https://www.mindnesthealth.com/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT03697837/Prot_SAP_000.pdf